CLINICAL TRIAL: NCT05383976
Title: A Feasibility Study to Improve Colorectal Cancer Screening Among Racially Diverse Zip Codes in a Persistent Poverty County Using Navigation and Machine Learning Predictive Algorithms
Brief Title: Improving Colorectal Cancer Screening in Racially Diverse Zip Codes Using Navigation and Machine Learning (PCSNaP)
Acronym: PCSNaP
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Principal Investigator, Carmen E. Guerra, MD, MSCE, FACP, Principle Investigator, Abramson Cancer Center at Penn Medicine
Other Study IDs: UPCC 09222; 850205 (Other: IRB)
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Results first posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2024-11

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Machine Learning Algorithms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients Residing in 18 zip codes in Western and Southwestern Philadelphia: The cohort will consist of patients residing in 18 zip codes in Western and Southwestern Philadelphia who have primary care providers in 4 Penn Medicine Internal Medicine practices and 3 Penn Medicine Family Medicine Practices.
  Interventions: Other: Machine Learning Algorithm with Existing Penn Medicine CRC Patient Navigation Program

INTERVENTIONS:
Other: Machine Learning Algorithm with Existing Penn Medicine CRC Patient Navigation Program — This intervention will utilize the existing Penn Medicine CRC patient navigation program. There will be a monthly list of patients with unfilled coloscopies provided, that are risk-stratified according to the machine learning algorithm and select high-risk criteria. The navigation team will prioritize timely outreach and navigation to high-risk patients according to a script that communicates risk.

SUMMARY:
The overarching goal of the "PCSNaP" Research Study is to support the Abramson Cancer Center (ACC) of the University of Pennsylvania in carrying out its mission to increase colorectal cancer (CRC) screening completion among high-risk individuals living in a persistent poverty county by designing, conducting, disseminating and evaluating an electronic health record-based automated identification program to target effective, culturally-sensitive CRC screening navigation to individuals who have not completed an ordered colonoscopy or fecal immunochemical test (FIT).

DETAILED DESCRIPTION:
Specifically, the goals of this study are to: 1) Adapt a previously validated electronic health record (EHR)-based machine learning algorithm to predict colorectal cancer (CRC) detection by retraining the model using data from patients seen in primary care clinics serving zip codes with a high proportion of racial and ethnic minorities living in Philadelphia County, a persistent poverty county; and 2) Implement and evaluate the feasibility and effectiveness of an algorithm-based CRC navigation program to increase colorectal cancer screening among patients in Philadelphia county who are at high risk of CRC and have uncompleted colonoscopies.

Together, these novel projects aim to be the first to combine use of machine learning algorithms and patient navigation to increase guideline-based cancer screening in order to reduce the burden of CRC among high-risk individuals living in a persistent poverty county through targeted, culturally-sensitive navigation that addresses social factors that prevent CRC screening.

ELIGIBILITY:
Inclusion Criteria:

* Patients residing in 18 zip codes in Western and Southwestern Philadelphia who have primary care providers in 4 Penn Medicine Internal Medicine practices and 3 Penn Medicine Family Medicine Practices
* Patients who have had a colonoscopy order placed in the past 6 months and have not scheduled, cancelled, or no-showed to their colonoscopy

Exclusion Criteria:

* Not applicable

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The cohort will consist of patients residing in 18 zip codes in Western and Southwestern Philadelphia who have primary care providers in 4 Penn Medicine Internal Medicine practices and 3 Penn Medicine Family Medicine Practices. Patients will have had a colonoscopy order placed in the past 6 months and have not scheduled, cancelled, or no-showed to their colonoscopy.
Sampling Method: Non-Probability Sample
Enrollment: 385 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Guerra, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Residing in 18 Zip Codes in Western and Southwestern Philadelphia: The cohort will consist of patients residing in 18 zip codes in Western and Southwestern Philadelphia who have primary care providers in 4 Penn Medicine Internal Medicine practices and 3 Penn Medicine Family Medicine Practices.
  Machine Learning Algorithm with Existing Penn Medicine CRC Patient Navigation Program: This intervention will utilize the existing Penn Medicine Colorectal Cancer patient navigation program. There will be a monthly list of patients with unfilled coloscopies provided, that are risk-stratified according to the machine learning algorithm and select high-risk criteria. The navigation team will prioritize timely outreach and navigation to high-risk patients according to a script that communicates risk.
- Controls: The cohort will consist of matched controls for the patients in the intervention cohort, also residing in the same 18 zip codes in Western and Southwestern Philadelphia with primary care providers in same 4 Penn Medicine Internal Medicine practices and 3 Penn Medicine Family Medicine Practices. Using clinical and sociodemographic characteristics, we will create matched cohorts of patients between the intervention participants and historical controls from the same clinics in the year prior.
Period: Overall Study
Arm/Group | Patients Residing in 18 Zip Codes in Western and Southwestern Philadelphia | Controls
Started | 201 | 184
Completed | 199 | 183
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients Residing in 18 Zip Codes in Western and Southwestern Philadelphia | Controls | Total
Number analyzed (Participants) | 201 | 184 | 385
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 135 | 145 | 280
  >=65 years | 66 | 39 | 105
Age, Continuous [Mean (Full Range); unit: years] | 61.28 [45 to 74] | 56.91 [45 to 73] | 59.10 [45 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 127 | 116 | 243
  Male | 74 | 68 | 142
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 16 | 34
  Not Hispanic or Latino | 183 | 168 | 351
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 134 | 134 | 268
  White | 34 | 29 | 63
  More than one race | 1 | 3 | 4
  Unknown or Not Reported | 29 | 13 | 42
Region of Enrollment [Number; unit: participants]
  United States | 201 | 184 | 385

OUTCOME MEASURES:

1. Primary Outcome: Enrollment in Navigator Program (Feasibility)
Description: Number of patients that participate in the navigation program
Time Frame: During the three month enrollment period
Population: Population consists of intervention patients who were correctly identified by the machine learning algorithm as needing to complete colorectal cancer screening and were eligible for navigation.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Residing in 18 Zip Codes in Western and Southwestern Philadelphia
Number analyzed (Participants) | 119
Participants | 79

2. Primary Outcome: Completion of Colorectal Cancer Screening
Description: Number of patients that have completed their colonoscopy or Fecal Immunochemical Test (FIT)
Time Frame: Within the three month enrollment period and three month follow-up period
Population: Population consists of intervention and control patients identified by the machine learning algorithm as needing to complete colorectal cancer screening.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Residing in 18 Zip Codes in Western and Southwestern Philadelphia | Controls
Number analyzed (Participants) | 199 | 183
Participants | 92 | 79

3. Primary Outcome: Number of Participants With Adenoma Detection
Description: Rate of adenomas after completion of colonoscopy
Time Frame: Within the three month enrollment period and three month follow-up period
Population: Population consists of patients who completed a colonoscopy during the study period.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients Residing in 18 Zip Codes in Western and Southwestern Philadelphia | Controls
Number analyzed (Participants) | 59 | 52
Participants | 21 | 15

ADVERSE EVENTS:
Time Frame: Adverse event data were not collected for this study.
Arm/Group | Patients Residing in 18 Zip Codes in Western and Southwestern Philadelphia | Controls
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-26): https://cdn.clinicaltrials.gov/large-docs/76/NCT05383976/Prot_SAP_000.pdf